CLINICAL TRIAL: NCT02924740
Title: The Effects of Vaginal Tampon Training Added to Pelvic Floor Muscle Training in Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gursen, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 16/506-18
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; quality of life; pelvic floor muscle training; pelvic floor muscle exercises; vaginal tampon training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): pelvic floor muscle training
  Interventions: Behavioral: Pelvic Floor Muscle Training
- intervention (Experimental): vaginal tampon training.
  Interventions: Behavioral: Pelvic Floor Muscle Training; Behavioral: Vaginal Tampon Training

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — Pelvic floor muscle training consist of fast (2 second) and slow contractions (5-s contraction, 10-s hold, 5-s relaxation, totally 20-s). One set of exercises includes ten fast and ten slow voluntary PFM contractions (VPFMCs). During week 1 and 2, participants will be instructed to perform two sets of exercises per day (20 fast and 20 slow contractions per day), which was progressively increased by two sets: four sets per day at week 3 and 4 (40 fast and 40 slow contractions per day); six sets per day at week 5 and 6 (60 fast and 60 slow contractions per day); eight sets per day at week 7 and 8 (80 fast and 80 slow contractions per day); ten sets per day from week 9 to week 12 (100 fast and 100 slow contractions per day).
Behavioral: Vaginal Tampon Training — Vaginal tampon training will be applied for 5 days a week for 12 weeks. Exercises with tampons will be performed two days a week by physiotherapist (first author) and three days a week by patients. One set of tampon exercises consist 15 contractions. During vaginal tampon training, from week 1 to week 12, patients were instructed to perform two sets of exercises for five days a week (two days by physiotherapist, three days by themselves).
  Arms: intervention

SUMMARY:
Pelvic Floor Muscle Training (PFMT) is the basis of conservative treatment in women with SUI. In systematic reviews, PFMT was recommended as a first option for treatment of SUI. The aim of PFMT is to improve sphincter activity and increase the support of bladder and urethra. Recommendations regarding the prevention and treatment of SUI with PFMT include Knack maneuver (the conscious contraction of the pelvic floor before and during the abdominal pressure increases); pelvic floor exercises to enhance the structural support and endurance of pelvic floor muscles; adding transversus abdominis contraction; and functional rehabilitation.It was reported that the progressive overload principle should be considered to improve the muscle strength and endurance. According to this principal, resistance against to movement, duration and/or frequency should be increased to obtain the optimal response. There are a lot of methods to run a muscle or muscle group based on the progressive overload principal. These are adding resistance or weight, increasing the duration and number of contraction, changing the type of exercise and the range of movement. In the literature, it was reported that special vaginal or rectal tools, vaginal cones or tampons might be used to establish resistance during the pelvic floor muscle exercises.the use of cones in a different way may provide extra benefit for patients: patients can be instructed to perform pelvic floor muscle contraction and try to pull the cone or the other tools out of the vagina. In this study, investigators preferred to use vaginal tampons since pulling the cone out of the vagina cause the elimination of the weight of the cone. Vaginal tampons are also sterile, hygienic, and single use. There is no study investigates the effects of vaginal tampon exercises in the literature. Therefore, the aim of this study is to investigate the effect of the vaginal tampon training adding to PFMT on symptoms of the urinary incontinence, the strength and the endurance of pelvic floor muscles and the quality of life.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is defined by the International Urogynecological Association and the International Continence Society (IUGA/ICS) as a complaint of involuntary loss of urine which is objectively shown and causing hygienic and social problems. Stress urinary incontinence (SUI) is defined as involuntary loss of urine on effort or physical exertion, or on sneezing or coughing. Pelvic Floor Muscle Training (PFMT) is the basis of conservative treatment in women with SUI. In systematic reviews, PFMT was recommended as a first option for treatment of SUI. The aim of PFMT is to improve sphincter activity and increase the support of bladder and urethra. Recommendations regarding the prevention and treatment of SUI with PFMT include Knack maneuver (the conscious contraction of the pelvic floor before and during the abdominal pressure increases); pelvic floor exercises to enhance the structural support and endurance of pelvic floor muscles; adding transversus abdominis contraction; and functional rehabilitation. It was reported that the progressive overload principle should be considered to improve the muscle strength and endurance. According to this principal, resistance against to movement, duration and/or frequency should be increased to obtain the optimal response. There are a lot of methods to run a muscle or muscle group based on the progressive overload principal. These are adding resistance or weight, increasing the duration and number of contraction, changing the type of exercise and the range of movement. In the literature, it was reported that special vaginal or rectal tools, vaginal cones or tampons might be used to establish resistance during the pelvic floor muscle exercises. It was found that the effect of exercises applying with a device was similar with PFMT in women with SUI and mixed type UI. Vaginal cones are weights that put into the vagina. The theory of the use of vaginal cones is that when the feeling of slipping is perceived, reflex or voluntary contraction of pelvic floor muscles occur to avoid this slipping. It was reported that the use of cones should be questioned in terms of exercise physiology. Holding the cone for 15-20 minutes may result in decreased blood supply, decreased oxygen consumption, muscle fatigue and pain, and contraction of other muscle. On the other hand, the use of cones in a different way may provide extra benefit for patients: patients can be instructed to perform pelvic floor muscle contraction and try to pull the cone or the other tools out of the vagina. In this study, investigators preferred to use vaginal tampons since pulling the cone out of the vagina cause the elimination of the weight of cone. Vaginal tampons are also sterile, hygienic, and single use. There is also no study investigates the effects of vaginal tampon exercises in the literature. Therefore, the aim of this study is to investigate the effect of the vaginal tampon training adding to PFMT on symptoms of the urinary incontinence, the strength and the endurance of pelvic floor muscles and the quality of life. Vaginal tampon training will be applied for 5 days a week for 12 weeks. Vaginal tampon exercises will be performed two days a week by physiotherapist (first author) and three days a week by patients. One set of tampon exercises consist 15 contractions. During vaginal tampon training, from week 1 to week 12, patients were instructed to perform two sets of exercises for five days a week (two days by physiotherapist, three days by themselves). Both groups will complete PFMT consisting of fast (2 second) and slow contractions (5-s contraction, 10-s hold, 5-s relaxation, totally 20-s). One set of exercises includes ten fast and ten slow voluntary PFM contractions (VPFMCs). During week 1 and 2, participants will be instructed to perform two sets of exercises per day (20 fast and 20 slow contractions per day), which was progressively increased by two sets: four sets per day at week 3 and 4 (40 fast and 40 slow contractions per day); six sets per day at week 5 and 6 (60 fast and 60 slow contractions per day); eight sets per day at week 7 and 8 (80 fast and 80 slow contractions per day); ten sets per day from week 9 to week 12 (100 fast and 100 slow contractions per day). Patients were advised to exercise while in the supine, seated, and upright positions and to integrate these exercises into their daily activities, e.g., while watching television, waiting for something, traveling.

ELIGIBILITY:
Inclusion Criteria:

* having symptoms of SUI according to MESA urinary incontinence questionnaire; age>18 and < 65 years; having the ability of pelvic floor muscle contraction, being free of UI medications for at least 4 weeks before the start of the study; and sufficient literacy to complete required forms and urinary diaries and perform training protocols.

Exclusion Criteria:

* antenatal or postnatal women (up to 3 months after delivery), women with persistent urinary tract infections, impaired mental state, Stage 3 and 4 pelvic organ prolapse (POP), neurological disorders, and who received concurrent or recent physiotherapy intervention (within the last year).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Global rating of improvement | change from baseline subjective improvement at 12 weeks
  A four-point scale (worse, unchanged, improved, cured) was used to determine the subjective perception of SUI improvement

SECONDARY OUTCOMES:
Pelvic floor muscle strength (PFMS) | change from baseline pelvic floor muscle strength at 12 weeks
  A vaginal perineometer (Cardio Design Pty Ltd., Australia) will be used to assess PFME with an arbitrary scale of 0-12.
Pelvic floor muscle endurance (PFME) | change from baseline pelvic floor muscle endurance at 12 weeks
  A vaginal perineometer (Cardio Design Pty Ltd., Australia) will be used to assess PFME with an arbitrary scale of 0-12.
Severity of urinary incontinence | change from baseline severity of incontinence at 12 weeks
  The severity of urinary incontinence will be questioned using the Incontinence Severity Index (ISI). The ISI included two items such as the frequency of urinary incontinence and amount of urinary incontinence. The total score is calculated by multiplying these items. The total score of ISI rages from 0 to 12. Higher scores presents severe urinary incontinence.
Frequency of micturition | change from baseline subjective improvement at 12 weeks
  Participants will complete three 24-h frequency volume charts on 3 nonconsecutive days, and the mean of the 3 days are obtained for analysis
Incontinent episodes | change from baseline incontinent episodes at 12 weeks
  Participants will complete three 24-h frequency volume charts on 3 nonconsecutive days, and the mean of the 3 days are obtained for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kashanian M, Ali SS, Nazemi M, Bahasadri S. Evaluation of the effect of pelvic floor muscle training (PFMT or Kegel exercise) and assisted pelvic floor muscle training (APFMT) by a resistance device (Kegelmaster device) on the urinary incontinence in women: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):218-23. doi: 10.1016/j.ejogrb.2011.06.037. Epub 2011 Jul 7. PMID 21741151
- [Background] Bump RC, Hurt WG, Fantl JA, Wyman JF. Assessment of Kegel pelvic muscle exercise performance after brief verbal instruction. Am J Obstet Gynecol. 1991 Aug;165(2):322-7; discussion 327-9. doi: 10.1016/0002-9378(91)90085-6. PMID 1872333
- [Background] Hay-Smith EJ, Bo Berghmans LC, Hendriks HJ, de Bie RA, van Waalwijk van Doorn ES. Pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2001;(1):CD001407. doi: 10.1002/14651858.CD001407. PMID 11279716
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Orhan C, Akbayrak T, Ozgul S, Baran E, Uzelpasaci E, Nakip G, Ozgul N, Beksac MS. Effects of vaginal tampon training added to pelvic floor muscle training in women with stress urinary incontinence: randomized controlled trial. Int Urogynecol J. 2019 Feb;30(2):219-229. doi: 10.1007/s00192-018-3585-7. Epub 2018 Mar 13. PMID 29536140